CLINICAL TRIAL: NCT06420076
Title: This is an Open, Single-arm, Clinical Study to Evaluate the Efficacy and Safety of Anti-CD7/CD5 CAR-T Cells in the Treatment of Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia (T-ALL), ETP-ALL, and Lymphoblastic Lymphoma (TLBL).
Brief Title: Sequential CAR-T Cells Therapy for CD5/CD7 Positive T-cell Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma Using CD5/CD7-Specific CAR-T Cells
Acronym: BAH246
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202496
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: T Cell Lymphoma; T Cell Leukemia; T-cell Acute Lymphoblastic Leukemia; T-Cell Lymphoma of CNS; T Cell Prolymphocytic Leukemia; T Cell Childhood ALL
Keywords: CAR-T; CD5; CD7; ETP-ALL
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, T-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic, T-Cell

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this clinical trial will receive a carefully designed treatment regimen. Prior to the infusion of CD5 and CD7 CAR-T cells, participants will undergo preconditioning chemotherapy. This chemotherapy serves to create an optimal environment for CAR-T cell therapy to effectively target and eliminate malignant B cells. Following chemotherapy, participants will receive the infusion of CD5 and CD7 CAR-T cells.
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential CAR-T Cells Targeting (CD5/CD7 CAR T cells, chemotherapy) (Experimental): Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive CD5/CD7 CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of CD5/CD7 CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of CD5/CD7 CAR T cells.
  Interventions: Biological: CD5/CD7 CAR-T

INTERVENTIONS:
Biological: CD5/CD7 CAR-T — The intervention in this clinical trial involves a novel approach using CD5/CD7 Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Patients in the trial will undergo the following regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  CD5/CD7 Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, CD5/CD7 CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial CD5/CD7 CAR-T cell infusion without unacceptable side effects and sufficient CAR-T cell availability may receive 2 or 3 additional doses.
  Other Names: EB-BH2026

SUMMARY:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. Besides CD19, many other molecules such as CD22, CD30,BCMA,CD123, etc. may be the potential to develop the corresponding CAR-T cells to treat patients whose tumors express those markers. In this study, investigators will evaluate the safety and efficacy of Sequential CAR-T Cells Targeting CD5/CD7 in patients with patients with relapsed or refractory T-ALL/LBL/ETP-ALL. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, disease status after treatment will also be evaluated.

DETAILED DESCRIPTION:
Acute lymphoblast leukemia (T-ALL) is a neoplastic lymphoid leukemia characterized by the proliferation of immature precursor T cells. The combined chemotherapy has significantly improved the prognosis of T-acute lymphoblast leukemia/lymphoma. However, once the disease appears to be relapsed/refractory, there are limited treatment options, and the overall prognosis is extremely poor. Therefore, exploring safe and effective treatments is a critical unmet medical need. The patients will receive Sequential CAR-T Cells Targeting CD5/CD7 to examine the safety and, possibly the efficacy of CD5 CAR T-Cells in CD5+ CD7+ relapsed or refractory acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent; Patients volunteer to participate in the clinical trial;
* Diagnosis is mainly based on the World Health Organization (WHO) 2008;
* Complete remission cannot be achieved after induction therapy; recurrence occurs after completion remission; the burden of leukemic blasts in the peripheral blood or bone marrow is greater than 5%;
* Leukemic blast cells express CD7/CD5 (CD7 OR CD5 positive by flow cytometry or immunohistochemistry ≥70%);
* The expected survival period is greater than 12 weeks;
* ECOG score ≤2;
* Age 2-60 years old;
* HGB≥70g/L (can be transfused);
* Total bilirubin does not exceed 3 times the upper limit of normal value, and AST and ALT do not exceed 5 times the upper limit of normal value.

Exclusion Criteria:

* Patients declining to consent for treatment
* Prior solid organ transplantation
* One of the following cardiac issues: atrial fibrillation; myocardial infarction within the past 12 months; prolonged QT syndrome or secondary QT prolongation; clinically significant pericardial effusion; cardiac insufficiency NYHA (New York Heart Association) III or IV;
* History of severe pulmonary dysfunction diseases;
* Severe infection or persistent infection cannot be effectively controlled;
* Severe autoimmune disease or congenital immunodeficiency;
* Active hepatitis;
* Human immunodeficiency virus (HIV) infection;
* Clinically significant viral infections, or uncontrollable viral reactivation, including EBV (Epstein-Barr virus).

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
The number and incidence of adverse events after CD7/CD5 CAR infusion. | 28 days
  Evaluation of all possible adverse reactions, including the number, incidence, and severity of symptoms such as cytokine release syndromes and neurotoxicity within 3 months after CAR-T infusion
Disease response to CD7/CD5 CAR T cells | 1 year
  The disease response to CD7/CD5 CAR T cells is evaluated by bone marrow biopsy and aspirate within 1 year after CAR infusion. The proportion of subjects receiving CD7/CD5 CAR T infusion to 1) morphological remission (blasts <5%): 2) flow cytometry analysis was blast negative, and 3) molecular biological remission (if applicable).

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided